CLINICAL TRIAL: NCT04578990
Title: Supervised Physical Activity in Subjects With Symptomatic Peripheral Arterial Disease. ARTPERfit Randomized Clinical Trial.
Brief Title: ARTPERfit Clinical Trial.
Acronym: ARTPERfit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI20/00129
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Arterial Disease; Arteriosclerosis
Keywords: Peripheral Arterial Disease; Physical Activity; Intermittent Claudication; Cardiovascular Disease; Ankle Brachial Index; Treadmill Test; Resistance Training; Functional Decline; Quality of Life
MeSH Terms: conditions — Peripheral Arterial Disease; Arteriosclerosis; Motor Activity; Intermittent Claudication; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized longitudinal controlled trial, parallel, blinded to the analysis, with a sample of participants studied between 3 and 6 months after starting a physical exercise program. Participants will be randomly assigned to four groups. Intervention walking group: The intervention will consist of carrying out the walking training progression. The strength group will carry out a resistance training program. The concurrent training intervention group will carry out an exercise program that will alternate strength and endurance training in the same session. Both experimental groups will hold 36-72 sessions, with a frequency of 3 sessions per week and 60 minutes per session. The control group will receive standard advice consisting of the recommendation to perform aerobic exercise at the lower limbs level warning.
Masking Description: Analysis masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Walking intervention group (Experimental): It will consist of performing the Treadmill training progression for 36-72 sessions. 3 sessions of 60 minutes, will be held weekly.
  Interventions: Other: Walking intervention
- Strength intervention group (Experimental): The training program consists of performing a training program with resistance exercises for 36-72 weeks.
  Interventions: Other: Strength intervention
- Concurrent intervention group (Experimental): The training program consists of alternating strength and resistance stimuli in the same session for 36-72 weeks. There will be 3 weekly sessions of 60 minutes, where exercises with resistance will be applied for 35 minutes and to complete the 60 minutes, the same guidelines will be followed as in the walking exercise, applying resistance stimuli.
  Interventions: Other: Concurrent intervention
- Control group (No Intervention): It will receive standard advice consisting of the recommendation to perform aerobic exercise at the lower limbs level.

INTERVENTIONS:
Other: Walking intervention — It will consist of performing the Treadmill training progression for 36-72 sessions. 3 sessions of 60 minutes, will be held weekly.
  Depending on the data obtained in Visit 1, the speed will be determined for each patient and the degree of the initial slope that is comfortable when walking until it induces symptoms of moderate intermittent claudication. The progression of the intensity of the speed and incline of the slope will be increased progressively and individually for each patient.
  Arms: Walking intervention group
Other: Strength intervention — The training program consists of performing a training program with resistance exercises for 36-72 weeks. There will be 3 weekly sessions of 60 minutes, where exercises with resistance will be applied. The same guidelines will be followed as in the walking exercise, but in this case, applying force stimuli. If symptoms of moderate intermittent claudication occur (3-4) based on the Claudication Symptom Rating Scale in 5-10 minutes, a period of rest (sitting or standing) will be performed until the pain disappears at the level of the lower limb. This sequence will be repeated until the strength training session is completed. The progression of force stimuli will be increased weekly depending on the subjective perception of the patient's effort and according to the guidelines set by our group of investigation.
  Arms: Strength intervention group
Other: Concurrent intervention — The training program consists of alternating strength and resistance stimuli in the same session for 36-72 weeks. There will be 3 weekly sessions of 60 minutes, where exercises with resistance will be applied for 35 minutes and to complete the 60 minutes, the same guidelines will be followed as in the walking exercise, applying resistance stimuli. If claudication symptoms occur moderate intermittent (3-4) based on the Claudication Symptom Rating Scale in 5-10 minutes, a period of rest (sitting or standing) will be performed until the pain in the lower extremity disappears. This sequence will be repeated until the 20 minutes established to end the session are completed concurrent training. The progression of the strength and resistance stimuli will be increased weekly depending on the perception subjective effort of the patient and according to the guidelines established by our research group.
  Arms: Concurrent intervention group

SUMMARY:
Peripheral arterial disease is part of the diseases derived from arteriosclerosis are the leading cause of mortality in developed countries. There is evidence of the benefits of physical exercise programs supervised in patients with cardiovascular risk. Despite being a treatment with proven efficacy and relatively inexpensive, it continues being little used for the management of patients with intermittent claudication caused by peripheral arterial disease.

The objective of this study is to develop an evidence-based intervention strategy on the effectiveness of supervised physical exercise in intermittent claudication to determine its impact compared to standard counselling in these patients.

DETAILED DESCRIPTION:
Peripheral arterial disease is part of the diseases derived from arteriosclerosis, such as myocardial infarction or stroke. These entities are the leading cause of mortality in developed countries. The peripheral arterial disease is a narrowing of the diameter of the arteries in the legs due to plaque formation of atheroma. When the obstruction is significant enough, there is a decrease in blood flow to the musculature of the lower limbs and consequently, depending on the severity of the narrowing, we can find from asymptomatic patients to patients with atrophic lesions, going through different degrees of pain when walking or at rest.

It is estimated that in 2010 more than 200 million people had peripheral arterial disease worldwide, with symptoms that range from mild to severe. The forecast is heading towards an increase in prevalence due to the increase in the life span of the world population and cardiovascular risk factors.

There is evidence in countries with high cardiovascular risk regarding the benefit obtained in physical exercise programs supervised in patients with pain when walking, both in increasing the distance walked and in prolonging at the time of onset of pain. Despite being a treatment with proven efficacy and relatively inexpensive, it continues being little used for the management of patients with intermittent claudication caused by arteriopathy in Spain.

This project aims to assess the effectiveness of various supervised physical exercise programs in patients with Symptomatic Peripheral Artery Disease (Intermittent Claudication) versus single advice to exercise without supervision. After a first initial assessment visit, four groups will be formed at random. A control group who will be given standard advice to perform physical exercise and three experimental intervention groups. They will be assessed at 3 and 6 months after performing sessions of supervised exercise lasting one hour 3 times a week and 12 months after the initial visit, (after 6 months of end supervised exercise sessions). The impact in terms of changes in quality of life will also be evaluated.

In the longer term, and depending on the results obtained, it is intended to implement a similar intervention, at the level of primary care, or as close as possible to the place of residence of this type of patient to facilitate the performance of the exercise, improve the symptoms and quality of life of these patients

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a peripheral arterial disease with symptoms of intermittent claudication
* Age> 40 years
* Signing of the informed consent to participate in the study

Exclusion Criteria:

* Critical ischemia and/or acute lower extremity ischemia
* Previous bilateral lower extremity revascularization.
* Lower limb amputation
* Major surgery in the previous 3 months or scheduled in the next year
* Cardiovascular, pulmonary, neurological and osteoarticular diseases that prevent the performance of the intervention.
* The appearance of intermittent claudication 30-45 minutes after the start of a claudication.
* Inability to go to the centre due to lack of time or limiting illness
* To participate, subjects must obtain medical consent to participate in a physical exercise intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain-free walking distance | 3 months from the start of the study
  Pain-free walking distance using Treadmill based walking
Pain-free walking distance | 6 months from the start of the study
  Pain-free walking distance using Treadmill based walking
Pain-free walking distance | 3 months from the start of the study
  Pain-free walking distance using the 6-minute walk test distance
Pain-free walking distance | 6 months from the start of the study
  Pain-free walking distance using the 6-minute walk test distance
General functional state | 3 months from the start of the study
  General functional state using the Barthel questionnaire.
General functional state | 6 months from the start of the study
  General functional state using the Barthel questionnaire.
Perceived quality of life level | 3 months from the start of the study
  Perceived quality of life level
Perceived quality of life level | 6 months from the start of the study
  Perceived quality of life level
Ankle-Brachial Index (ABI) | 3 months from the start of the study
  To know if the proposed training programs improve the ankle-brachial index.
Ankle-Brachial Index (ABI) | 6 months from the start of the study
  To know if the proposed training programs improve the ankle-brachial index.

SECONDARY OUTCOMES:
Maintenance of objective in the long term | 12 months from the start of the study
  Determine the maintenance of objectives 1, 2 and 3, 6 months after completing the intervention
Keep exercising in the long term | 12 months from the start of the study
  To know the proportion of subjects who continue to exercise 6 months after completing the study
Severity of peripheral arterial disease | 3 and 6 months from the start of the study
  Determine objectives 1, 2 and 3 concerning the severity of peripheral arterial disease (according to baseline ABI) at 3 and 6 months of an exercise program supervised physicist.
Ankle-Brachial Index in the long term | 12 months from the start of the study
  Analyze the changes in the ankle-brachial index at 12 months from the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Alzamora Sas, MD and PhD, Principal Investigator — Institut Català de la Salut
Locations (1):
- Unitat de Suport a la Recerca (Metropolitana Nord), Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Felix-Redondo FJ, Fernandez-Berges D, Grau M, Baena-Diez JM, Mostaza JM, Vila J. Prevalence and clinical characteristics of peripheral arterial disease in the study population Hermex. Rev Esp Cardiol (Engl Ed). 2012 Aug;65(8):726-33. doi: 10.1016/j.recesp.2012.03.008. Epub 2012 Jun 22. English, Spanish. PMID 22727799
- [Background] Ramos R, Quesada M, Solanas P, Subirana I, Sala J, Vila J, Masia R, Cerezo C, Elosua R, Grau M, Cordon F, Juvinya D, Fito M, Isabel Covas M, Clara A, Angel Munoz M, Marrugat J; REGICOR Investigators. Prevalence of symptomatic and asymptomatic peripheral arterial disease and the value of the ankle-brachial index to stratify cardiovascular risk. Eur J Vasc Endovasc Surg. 2009 Sep;38(3):305-11. doi: 10.1016/j.ejvs.2009.04.013. Epub 2009 Jun 10. PMID 19515589
- [Background] Alzamora MT, Fores R, Baena-Diez JM, Pera G, Toran P, Sorribes M, Vicheto M, Reina MD, Sancho A, Albaladejo C, Llussa J; PERART/ARTPER study group. The peripheral arterial disease study (PERART/ARTPER): prevalence and risk factors in the general population. BMC Public Health. 2010 Jan 27;10:38. doi: 10.1186/1471-2458-10-38. PMID 20529387
- [Background] Blanes JI, Cairols MA, Marrugat J; ESTIME. Prevalence of peripheral artery disease and its associated risk factors in Spain: The ESTIME Study. Int Angiol. 2009 Feb;28(1):20-5. PMID 19190551
- [Background] Sampson UK, Fowkes FG, McDermott MM, Criqui MH, Aboyans V, Norman PE, Forouzanfar MH, Naghavi M, Song Y, Harrell FE Jr, Denenberg JO, Mensah GA, Ezzati M, Murray C. Global and regional burden of death and disability from peripheral artery disease: 21 world regions, 1990 to 2010. Glob Heart. 2014 Mar;9(1):145-158.e21. doi: 10.1016/j.gheart.2013.12.008. PMID 25432124
- [Background] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Background] Alzamora MT, Fores R, Pera G, Toran P, Heras A, Sorribes M, Baena-Diez JM, Urrea M, Alegre J, Viozquez M, Vela C. Ankle-brachial index and the incidence of cardiovascular events in the Mediterranean low cardiovascular risk population ARTPER cohort. BMC Cardiovasc Disord. 2013 Dec 17;13:119. doi: 10.1186/1471-2261-13-119. PMID 24341531
- [Background] Criqui MH, McClelland RL, McDermott MM, Allison MA, Blumenthal RS, Aboyans V, Ix JH, Burke GL, Liu K, Shea S. The ankle-brachial index and incident cardiovascular events in the MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2010 Oct 26;56(18):1506-12. doi: 10.1016/j.jacc.2010.04.060. PMID 20951328
- [Background] Mostaza JM, Puras E, Blasco M, Lahoz C, Samaniego ML. Utilization of evidence-based cardiovascular therapies and achievement of therapeutic goals in patients with peripheral artery disease. Rev Esp Cardiol (Engl Ed). 2012 Aug;65(8):713-8. doi: 10.1016/j.recesp.2012.02.020. Epub 2012 May 31. English, Spanish. PMID 22658690
- [Background] Fores R, Alzamora MT, Pera G, Valverde M, Angla M, Baena-Diez JM, Mundet-Tuduri X. Evolution and degree of control of cardiovascular risk factors after 5 years of follow-up and their relationship with the incidence of peripheral arterial disease: ARTPER cohort. Med Clin (Barc). 2017 Feb 9;148(3):107-113. doi: 10.1016/j.medcli.2016.09.043. Epub 2016 Nov 25. English, Spanish. PMID 27894602
- [Background] Marrett E, DiBonaventura Md, Zhang Q. Burden of peripheral arterial disease in Europe and the United States: a patient survey. Health Qual Life Outcomes. 2013 Oct 22;11:175. doi: 10.1186/1477-7525-11-175. PMID 24148832
- [Background] Regensteiner JG, Hiatt WR, Coll JR, Criqui MH, Treat-Jacobson D, McDermott MM, Hirsch AT. The impact of peripheral arterial disease on health-related quality of life in the Peripheral Arterial Disease Awareness, Risk, and Treatment: New Resources for Survival (PARTNERS) Program. Vasc Med. 2008 Feb;13(1):15-24. doi: 10.1177/1358863X07084911. PMID 18372434
- [Background] McDermott MM, Greenland P, Liu K, Guralnik JM, Criqui MH, Dolan NC, Chan C, Celic L, Pearce WH, Schneider JR, Sharma L, Clark E, Gibson D, Martin GJ. Leg symptoms in peripheral arterial disease: associated clinical characteristics and functional impairment. JAMA. 2001 Oct 3;286(13):1599-606. doi: 10.1001/jama.286.13.1599. PMID 11585483
- [Background] McDermott MM, Liu K, Greenland P, Guralnik JM, Criqui MH, Chan C, Pearce WH, Schneider JR, Ferrucci L, Celic L, Taylor LM, Vonesh E, Martin GJ, Clark E. Functional decline in peripheral arterial disease: associations with the ankle brachial index and leg symptoms. JAMA. 2004 Jul 28;292(4):453-61. doi: 10.1001/jama.292.4.453. PMID 15280343
- [Background] F.S.Lozano Sánchez, J.R March García E Carrasco Carrasco. Profile of patients with intermittent claudication in Spain. The VITAL Study. Angiologia. 2013;65:131-140
- [Background] Frank U, Nikol S, Belch J, Boc V, Brodmann M, Carpentier PH, Chraim A, Canning C, Dimakakos E, Gottsater A, Heiss C, Mazzolai L, Madaric J, Olinic DM, Pecsvarady Z, Poredos P, Quere I, Roztocil K, Stanek A, Vasic D, Visona A, Wautrecht JC, Bulvas M, Colgan MP, Dorigo W, Houston G, Kahan T, Lawall H, Lindstedt I, Mahe G, Martini R, Pernod G, Przywara S, Righini M, Schlager O, Terlecki P. ESVM Guideline on peripheral arterial disease. Vasa. 2019 Sep;48(Suppl 102):1-79. doi: 10.1024/0301-1526/a000834. No abstract available. PMID 31789115
- [Background] Fowkes FG, Housley E, Cawood EH, Macintyre CC, Ruckley CV, Prescott RJ. Edinburgh Artery Study: prevalence of asymptomatic and symptomatic peripheral arterial disease in the general population. Int J Epidemiol. 1991 Jun;20(2):384-92. doi: 10.1093/ije/20.2.384. PMID 1917239
- [Background] Diehm C, Schuster A, Allenberg JR, Darius H, Haberl R, Lange S, Pittrow D, von Stritzky B, Tepohl G, Trampisch HJ. High prevalence of peripheral arterial disease and co-morbidity in 6880 primary care patients: cross-sectional study. Atherosclerosis. 2004 Jan;172(1):95-105. doi: 10.1016/s0021-9150(03)00204-1. PMID 14709362
- [Background] Vouyouka AG, Egorova NN, Salloum A, Kleinman L, Marin M, Faries PL, Moscowitz A. Lessons learned from the analysis of gender effect on risk factors and procedural outcomes of lower extremity arterial disease. J Vasc Surg. 2010 Nov;52(5):1196-202. doi: 10.1016/j.jvs.2010.05.106. Epub 2010 Jul 31. PMID 20674247
- [Background] Gallagher KA, Meltzer AJ, Ravin RA, Graham A, Connolly P, Escobar G, Shrikhande G, McKinsey JF. Gender differences in outcomes of endovascular treatment of infrainguinal peripheral artery disease. Vasc Endovascular Surg. 2011 Nov;45(8):703-11. doi: 10.1177/1538574411418008. Epub 2011 Sep 13. PMID 21914680
- [Background] Lane R, Harwood A, Watson L, Leng GC. Exercise for intermittent claudication. Cochrane Database Syst Rev. 2017 Dec 26;12(12):CD000990. doi: 10.1002/14651858.CD000990.pub4. PMID 29278423
- [Background] Vemulapalli S, Dolor RJ, Hasselblad V, Schmit K, Banks A, Heidenfelder B, Patel MR, Jones WS. Supervised vs unsupervised exercise for intermittent claudication: A systematic review and meta-analysis. Am Heart J. 2015 Jun;169(6):924-937.e3. doi: 10.1016/j.ahj.2015.03.009. Epub 2015 Mar 26. PMID 26027632
- [Background] Ahimastos AA, Pappas EP, Buttner PG, Walker PJ, Kingwell BA, Golledge J. A meta-analysis of the outcome of endovascular and noninvasive therapies in the treatment of intermittent claudication. J Vasc Surg. 2011 Nov;54(5):1511-21. doi: 10.1016/j.jvs.2011.06.106. Epub 2011 Sep 29. PMID 21958561
- [Background] Tunstall-Pedoe H, Kuulasmaa K, Amouyel P, Arveiler D, Rajakangas AM, Pajak A. Myocardial infarction and coronary deaths in the World Health Organization MONICA Project. Registration procedures, event rates, and case-fatality rates in 38 populations from 21 countries in four continents. Circulation. 1994 Jul;90(1):583-612. doi: 10.1161/01.cir.90.1.583. PMID 8026046
- [Background] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Background] McGuigan MR, Bronks R, Newton RU, Sharman MJ, Graham JC, Cody DV, Kraemer WJ. Resistance training in patients with peripheral arterial disease: effects on myosin isoforms, fiber type distribution, and capillary supply to skeletal muscle. J Gerontol A Biol Sci Med Sci. 2001 Jul;56(7):B302-10. doi: 10.1093/gerona/56.7.b302. PMID 11445595
- [Background] Mosti MP, Wang E, Wiggen ON, Helgerud J, Hoff J. Concurrent strength and endurance training improves physical capacity in patients with peripheral arterial disease. Scand J Med Sci Sports. 2011 Dec;21(6):e308-14. doi: 10.1111/j.1600-0838.2011.01294.x. Epub 2011 Mar 16. PMID 21410546
- [Background] Ferrieres J. The French paradox: lessons for other countries. Heart. 2004 Jan;90(1):107-11. doi: 10.1136/heart.90.1.107. No abstract available. PMID 14676260
- [Derived] Alzamora MT, Fores R, Serra N, Martinez E, Pera G, Seda G, Lopez Palencia J, Gomis M, Heras Tebar A, Valverde M, Garnacho MV, Toran P. Supervised physical activity in patients with symptomatic peripheral arterial disease: protocol for a randomized clinical trial (ARTPERfit Study). BMJ Open. 2022 Apr 27;12(4):e054352. doi: 10.1136/bmjopen-2021-054352. PMID 35477870